CLINICAL TRIAL: NCT04707287
Title: Association of Tumour Grade and Sex Steroid Receptor as a Prognostic Index in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Fazila Hashmi, Assistant Professor, Liaquat University of Medical & Health Sciences
Other Study IDs: LUMHS/REC/-17
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Sex steroid receptors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: All the patients irrespective of age, ethnicity and stage of disease will be including once the disease is confirmed after triple assessment
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention used. This is observational study

SUMMARY:
Null hypothesis: Histological grade of tumour bears no relation with the status of sex hormone receptors.

Alternate hypothesis: Both the histological grade of tumour and expression of sex steroid receptors are directly related to each other The investigators aim to;

1. see the relationship of sex steroid receptors with the histological grade of breast cancer.
2. evaluate the efficacy of steroid receptors as a prognostic factor

DETAILED DESCRIPTION:
Breast cancer accounts for the largest number of deaths amongst the female population worldwide. It is now considered as a systemic disease even if diagnosed at an initial stage, as the clinical behaviour cannot be accurately predicted. Due to this reason, it is subjected to new dimensions of research every day. The aggressiveness of the cancer is directly proportional to the histopathological grade at the time of diagnosis. This is true with reference to the clinical stage at the time of presentation, the probability to metastasize and potential to recur. The idea of steroids receptor expression by the tumour is not new, and to evaluate their status prior to the induction of hormone therapy is a must.

The sex steroids, which are produced intratumorally, include estrogen, progesterone, and androgens. They act on their specific receptors present on the cell surface, within the cytoplasm and at the nuclear membrane. It is a measurement of these receptors that decide the potential of an individual to respond to different types of hormones like estrogen receptor blockers and aromatase inhibitors. Do the histological grade of tumour bears some relation with the status of these receptors and can investigators predict and rely just on the cellular behaviour of tumour for the purpose of prognosis is still under investigation. This study is designed to see the relationship between the histopathological grade of the tumour with the expression of sex steroid receptors. It will also try to evaluate whether these receptors bear some prognostic value or not.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with breast cancer irrespective of age, gender and clinical stage

Exclusion Criteria:

* Any patient who lost to follow up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients irrespective of age, gender and stage of disease will be including once the disease is confirmed after triple assessment. We shall cover the population in the southern part of Pakistan.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Histopathology of tumour | 6 months
  The incidence of grade and type of breast cancer at the time of study will be recorded and analysed
Steroid receptor status | 6 months
  The concentrations of estrogen and progesterone receptor will be calculated and analysed.

SECONDARY OUTCOMES:
Age | 6 months
  The age of patient will be calculated and compared to the primary outcomes.
State of menstruation | 6 months
  The onset of premenopausal and postmenopausal status of patient will be recorded
Stage of tumour | 6 months
  The status of clinical and pathological stage of the breast cancer at the time of study will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Fazila Hashmi, Principal Investigator — Liaquat University of Medical and Health Sciences Jamshoro Pakistan
Locations (2):
- Pakistan (2):
  - Fazila Hashmi, Jāmshoro, Sindh
  - Liaquat University of Medical and Health Sciences, Jāmshoro

IPD SHARING:
Plan to Share IPD: Undecided
At the moment the facility is undecided about the plans to share the data

REFERENCES:
- [Background] Gadducci A, Biglia N, Sismondi P, Genazzani AR. Breast cancer and sex steroids: critical review of epidemiological, experimental and clinical investigations on etiopathogenesis, chemoprevention and endocrine treatment of breast cancer. Gynecol Endocrinol. 2005 Jun;20(6):343-60. doi: 10.1080/09513590500128492. PMID 16019385
- [Background] Folkerd E, Dowsett M. Sex hormones and breast cancer risk and prognosis. Breast. 2013 Aug;22 Suppl 2:S38-43. doi: 10.1016/j.breast.2013.07.007. PMID 24074790
- [Background] Gambardella A, Esposito D, Accardo G, Taddeo M, Letizia A, Tagliafierro R, Esposito K, Pasquali D. Sexual function and sex hormones in breast cancer patients. Endocrine. 2018 Jun;60(3):510-515. doi: 10.1007/s12020-017-1470-7. Epub 2017 Nov 14. PMID 29138989
- [Background] Stute P, Wildt L, Neulen J. The impact of micronized progesterone on breast cancer risk: a systematic review. Climacteric. 2018 Apr;21(2):111-122. doi: 10.1080/13697137.2017.1421925. Epub 2018 Jan 31. PMID 29384406
- [Background] Clendenen TV, Ge W, Koenig KL, Afanasyeva Y, Agnoli C, Brinton LA, Darvishian F, Dorgan JF, Eliassen AH, Falk RT, Hallmans G, Hankinson SE, Hoffman-Bolton J, Key TJ, Krogh V, Nichols HB, Sandler DP, Schoemaker MJ, Sluss PM, Sund M, Swerdlow AJ, Visvanathan K, Zeleniuch-Jacquotte A, Liu M. Breast cancer risk prediction in women aged 35-50 years: impact of including sex hormone concentrations in the Gail model. Breast Cancer Res. 2019 Mar 19;21(1):42. doi: 10.1186/s13058-019-1126-z. PMID 30890167